CLINICAL TRIAL: NCT04606602
Title: A Randomised, Double-blind, Placebo Controlled, First-in-human Study to Investigate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Response of SLN360 in Subjects With Elevated Lipoprotein(a)
Brief Title: Study to Investigate Safety, Tolerability, PK and PD Response of SLN360 in Subjects With Elevated Lipoprotein(a)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Silence Therapeutics plc (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SLN360-001
Record Dates: First submitted 2020-10-07; First posted 2020-10-28 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Hyperlipidemias; Dyslipidemias; Elevated Lp(a)
Keywords: Dyslipidemia, Dyslipoproteinemia, Hyperlipidemia, Hyperlipoproteinemia, Hyperlipoproteinemia (a), Lipoprotein, Lipoprotein (a)
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias; Hyperlipoproteinemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- 30 mg (Experimental)
  Interventions: Drug: SLN360
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 100 mg (Experimental)
  Interventions: Drug: SLN360
- 300 mg (Experimental)
  Interventions: Drug: SLN360
- 600 mg (Experimental)
  Interventions: Drug: SLN360
- 900 mg (Experimental)
  Interventions: Drug: SLN360
- 100 mg multi dose (Experimental)
  Interventions: Drug: SLN360
- 200 mg multi dose (Experimental)
  Interventions: Drug: SLN360
- 300 mg multi dose (Experimental)
  Interventions: Drug: SLN360
- 600 mg multi dose (Experimental)
  Interventions: Drug: SLN360
- Placebo multi dose (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLN360 — SLN360 for subcutaneous (s.c.) injection
  Arms: 100 mg; 100 mg multi dose; 200 mg multi dose; 30 mg; 300 mg; 300 mg multi dose; 600 mg; 600 mg multi dose; 900 mg
Drug: Placebo — Sodium chloride for subcutaneous (s.c.) injection
  Arms: Placebo; Placebo multi dose

SUMMARY:
This study will investigate the safety and tolerability of SLN360 in patients with elevated Lp(a).

DETAILED DESCRIPTION:
This first-in-human (FIH) study will investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of SLN360 after single ascending s.c. doses and multiple doses in healthy male and female subjects.

Up to 9 cohorts of 88 patients with elevated Lp(a) will be enrolled. Each patient will receive single or multiple doses of SLN360 or placebo given by subcutaneous (s.c) injection.

ELIGIBILITY:
Inclusion criteria:

* Elevated plasma Lp(a) ≥ 150nmol/L.
* All subjects must agree to adhere to appropriate contraception requirements.
* Subjects must provide written informed consent and be able to comply with all study requirements.
* Body mass index of ≥ 18 kg/m2 and ≤ 45 kg/m2.
* For the MD part: confirmed history of stable atherosclerortic cardiovascular disease.

Exclusion criteria:

* Single Ascending Dose only: any history of clinically overt cardiovascular disease, defined as acute coronary syndromes, myocardial infarction, stable angina, coronary or other revascularization, ischemic stroke or transient ischemic attack and atherosclerotic peripheral arterial disease.
* Multiple Dose only: recent history of acute cardiovascular disease events within 6 months of screening (including, but not limited to, acute myocardial infarction, unstable angina, acute stroke and acute limb ischemia).
* Moderate or severe hepatic cirrhosis with Child-Pugh grade B or C, or other current or previous liver disease.
* Active serious mental illness or psychiatric disorder, including but not limited to schizophrenia, bipolar disorder, or severe depression requiring current pharmacological intervention.
* Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrolment in the study or could interfere with the subject's participation in, or completion of the study.
* Subjects with previous or current use of medication or therapies significantly affecting Lp(a) level or hormone replacement therapy, unless on a stable dose for ≥ 8 weeks prior to screening
* History or clinical evidence of alcohol or illegal drug misuse within the 6 months before screening.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc, or intolerance to s.c. injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 150
  safety and tolerability will be reported separately following single-dose administration.
Incidence of treatment-emergent adverse events | Day 201
  safety and tolerability will be reported separately following multiple-dose administration.

SECONDARY OUTCOMES:
Pharmacokinetic: peak plasma concentration (Cmax) | Day 150 and Day 201
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.
Pharmacokinetic: area under the plasma concentration (AUC) | Day 150 and Day 201
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.
Pharmacokinetic: apparent total clearance from plasma after s.c injection (CL/F) | Day 150 and Day 201
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.
Pharmacodynamic: Change in Lp(a) | Day 150 and Day 201
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Jacksonville Center for Clinical Research Ltd., Jacksonville, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
- Australia (2):
  - Linear Clinical Research, Perth, Western Australia
  - Monash Medical Centre, Clayton
- Amsterdam Medical Centre, Amsterdam, Netherlands
- Hammersmith Medicines Research, London, United Kingdom

REFERENCES:
- [Result] Nissen SE, Wolski K, Balog C, Swerdlow DI, Scrimgeour AC, Rambaran C, Wilson RJ, Boyce M, Ray KK, Cho L, Watts GF, Koren M, Turner T, Stroes ES, Melgaard C, Campion GV. Single Ascending Dose Study of a Short Interfering RNA Targeting Lipoprotein(a) Production in Individuals With Elevated Plasma Lipoprotein(a) Levels. JAMA. 2022 May 3;327(17):1679-1687. doi: 10.1001/jama.2022.5050. PMID 35368052
- [Result] Nissen SE, Wolski K, Watts GF, Koren MJ, Fok H, Nicholls SJ, Rider DA, Cho L, Romano S, Melgaard C, Rambaran C. Single Ascending and Multiple-Dose Trial of Zerlasiran, a Short Interfering RNA Targeting Lipoprotein(a): A Randomized Clinical Trial. JAMA. 2024 May 14;331(18):1534-1543. doi: 10.1001/jama.2024.4504. PMID 38587822